CLINICAL TRIAL: NCT04886557
Title: Retrospective Image Analysis of Degenerative Lumbar Disease Patients
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-10-008BC
Record Dates: First submitted 2021-05-12; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Lumbar Spondylolisthesis
Keywords: Dynesys dynamic stabilization, range of motion
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DDS fixation: Adult patients with degenerative spondylolisthesis over L4-L5 received DDS with a minimum of 2-year follow-up were reviewed. Surgical indications were patients who failed to respond to conservative treatment for at least 6 months. The exclusion criteria were: (1) presence of degenerative scoliosis or spinal deformity, (2) prior spine surgery, (3) lost to follow-up, or (4) failure to complete the questionnaires or radiographic examinations.
  Interventions: Procedure: L4-L5 decompression and dynamic instrumentation

INTERVENTIONS:
Procedure: L4-L5 decompression and dynamic instrumentation — All surgeries were performed by a senior surgeon using a traditional midline approach. Stability-preserving lumbar decompression with facet joint undercutting was performed to preserve the facet joints as much as possible. In cases of severe stenosis, a bilateral partial facetectomy (< 25%) was performed for adequate decompression. Posterior tension of the supra- and inter-spinous ligaments was preserved at the most cranial level. Patients were encouraged to ambulate after drain removal and wear a soft lumbar orthosis for at least 3 months after the operation.

SUMMARY:
The Dynesys dynamic stabilization (DDS) system is considered a motion-preserving device. However, studies addressing the change in the range of motion (ROM) are limited. Therefore, this study aimed to investigate the factors influencing ROM change at the index surgical level, supra-index level, and whole lumbar spine, in addition to the association between ROM preservation and the incidence of screw-loosening.

DETAILED DESCRIPTION:
Decompression with instrumented fusion is an effective surgical intervention for lumbar degenerative spondylolisthesis with spinal stenosis. However, the range of motion (ROM) decreased at the index surgical level may lead to an increased ROM at the non-surgical level, increase biomechanical stress at the transitional adjacent segment, and lead to adjacent segment degeneration (ASD) .

The Dynesys dynamic stabilization (DDS) system is a pedicle screw-based, motion-preserving, and non-fusion stabilization developed as an alternative to the rigid instrumented fusion for degenerative spondylolisthesis. The aim of the DDS is to maintain segmental motion at index levels and to reduce the incidence of ASD. However, the actual impact of ROM has remained elusive. Prior studies have reported an average ROM loss of 1.1º to 17.3º 7 at index surgical level at an average of 24 months follow-up.

The change of ROM at index surgical, supra-index, and whole lumbar spine following DDS remains unclear. This study aims to investigate the factors influencing the ROM change at index surgical level, supra-index level, and whole lumbar spine, and the association between ROM preservation and the incidence of screw-loosening.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Diagnosed with degenerative spondylolisthesis over L4-L5
* Received DDS
* Received a minimum of 2-year follow-up were reviewed.

Exclusion Criteria:

* presence of degenerative scoliosis or spinal deformity,
* prior spine surgery,
* lost to follow-up, or
* failure to complete the questionnaires or radiographic examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with degenerative spondylolisthesis over L4-L5 who failed to respond to conservative treatment for at least 6 months and received Dynesys instrumentation.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Range of motion | All patients completed the follow-up assessment at postoperative 1-, 2-, 3-, 6-, 12-, and 24-months.
  The ROM change at index surgical level, supra-index level, and whole lumbar spine in degenerative lumbar diseased patients received dynesys dynamic instrumentation

SECONDARY OUTCOMES:
Screw loosening | All patients completed the follow-up assessment at postoperative 1-, 2-, 3-, 6-, 12-, and 24-months.
  Radiographic screw-loosening was defined as presence of a halo or double-halo sign on plain x-ray films

CONTACTS AND LOCATIONS:
Locations (1):
- Dep. of Orthopedics and Traumatology, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] St-Pierre GH, Jack A, Siddiqui MM, Henderson RL, Nataraj A. Nonfusion Does Not Prevent Adjacent Segment Disease: Dynesys Long-term Outcomes With Minimum Five-year Follow-up. Spine (Phila Pa 1976). 2016 Feb;41(3):265-73. doi: 10.1097/BRS.0000000000001158. PMID 26335675